CLINICAL TRIAL: NCT04403217
Title: Effect of MEDiterranean Diet on the microBIOME of Individuals With Type 2 Diabetes
Acronym: MEDBIOME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDBIOME
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes
Keywords: Gut microbiota; Mediterranean diet; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized structured dietary plan based on MD (Experimental): Participants will follow an individualized structured dietary plan based on Mediterranean diet for 12 weeks
  Interventions: Other: Individualized structured dietary plan based on MD

INTERVENTIONS:
Other: Individualized structured dietary plan based on MD — Participants will follow an individualized structured dietary plan based on Mediterranean diet for 12 weeks

SUMMARY:
Dysbiosis of gut microbiota is associated with the pathophysiology of type 2 diabetes. Mediterranean diet has been indicated as a dietary pattern that promote the integrity of gut barrier and that has positive impact in the metabolic control of subjects with type 2 diabetes. This is a 12-week, single-arm clinical study that aims to evaluate if the effect of Mediterranean diet in metabolic control of these subjects is mediated by gut microbiota. Subjects will receive personalized nutrition counseling where Mediterranean diet will be promoted.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with type 2 diabetes mellitus, according to the American Diabetes Association criteria;
* Ages 40-80 years;
* Non-smoker;
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Diabetes diagnosed before 40 years old;
* Changes in oral glycaemic-control medications in the last 3 months;
* Subjects with HbA1c levels under 6.4% or above 10%;
* Subjects under insulinotherapy;
* Subjects under corticotherapy;
* Subjects with triglycerides levels above 4.52 nmol/L (400 mg/dL);
* Intake of antibiotics in the last 12 weeks;
* Subjects with a diagnosis of any digestive disease including functional bowel disorders such as IBS.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in intestinal microbiota from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2) and 12-week post Mediterranean diet intervention (visit 3)
  Bacterial DNA will be extracted from fecal samples. 16SRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage
Changes in HbA1c levels (percent) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in HOMA-IR from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in HOMA-B (percent) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in HOMA-S (percent) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in fasting capillary blood glucose (mg/dL) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in fasting insulin (μU/mL) levels from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)

SECONDARY OUTCOMES:
Changes in diet quality from baseline to visit 3 | 1-week post run-in period (baseline), 12-week post Mediterranean diet intervention (visit 3)
  Mediterranean diet adherence will be evaluated using the Mediterranean Diet Adherence Screener (MEDAS) from the PREvención com Dieta MEDiterránea (PREDIMED) study. Responses that are favorable to the adoption of the Mediterranean diet are scored as 1 point, while responses that are unfavorable are scored as 0.
  The final score ranged between 0 and 14 and a MEDAS score greater than 9 indicates high adherence to the Mediterranean diet.
Changes in food intake from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
  3 non-consecutive 24-h dietary food recall using a photographic manual for food quantification
Changes in fasting serum total cholesterol (mg/dL) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in fasting serum high-density lipoprotein (HDL) (mg/dL) cholesterol from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in fasting serum low-density lipoprotein (LDL) (mg/dL) cholesterol from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in fasting serum triglycerides (mg/dL) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in total body fat mass (kg) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in free fat mass (kg) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)
Changes in waist perimeter (cm) from baseline to visit 2 and 3 | 1-week post run-in period (baseline), 4-week post Mediterranean diet intervention (visit 2), 12-week post Mediterranean diet intervention (visit 3)

CONTACTS AND LOCATIONS:
Locations (1):
- NOVA Medical School|Faculdade de Ciências Médicas, Universidade NOVA de Lisboa, Lisbon, Portugal